CLINICAL TRIAL: NCT02415413
Title: A Phase II Multicenter Study of Carfilzomib, Lenalidomide and Dexamethasone (KRd) as Induction Therapy, Followed by High-dose Therapy With Melphalan and Autologous Peripheral Blood Stem Cell Transplantation, Consolidation With KRd, and Maintenance With Lenalidomide and Dexamethasone in Patients ≤ 70 Years Old With Smoldering Multiple Myeloma (SMM) With High Risk of Progression to Symptomatic Myeloma
Brief Title: Carfilzomib in Treatment Patients Under 65 Years With High Risk Smoldering Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Celgene Corporation (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-CESAR
Record Dates: First submitted 2015-03-29; First posted 2015-04-14 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Smoldering Multiple Myeloma
Keywords: Smoldering multiple myeloma; Carfilzomib; Lenalidomide; Melphalan; Dexamethasone; Autologous stem cell transplantation
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carlizomib lenalidomide and low dose dexamethasone (Experimental): Induction treatment: patients included in the trial will receive an induction treatment for approximately 6 months (6 cycles of carfilzomib, lenalidomide and low dose dexamethasone (KRd)). After the third cycle of KRd, all patients will be mobilized with colony stimulating factor (G-CSF) alone to collect peripheral blood stem cell for the ASCT.
  High dose therapy followed by autologous stem cell transplantation: patients will receive melphalan 200 mg/m2 via intravenous followed by autologous stem cell transplantation (HDT-ASCT).
  Consolidation treatment: approximately 3 months after the autologous stem cell transplantation, patients will receive consolidation treatment for 2 months (2 cycles of carfilzomib, lenalidomide and low dose dexamethasone (KRd)).
  Maintenance treatment: subsequently they will start a maintenance treatment that will be administered for approximately 24 months (24 cycles of lenalidomide and low dose dexamethasone
  Interventions: Drug: carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Melphalan

INTERVENTIONS:
Drug: carfilzomib
Drug: Lenalidomide
Drug: Dexamethasone
Drug: Melphalan

SUMMARY:
Patients included in the study will receive induction treatment during 6 months, followed by receive high-dose therapy followed by peripheral blood stem cell transplantation.

Approximately 3 months after peripheral blood stem cell transplantation patients will receive consolidation treatment during 2 months.

Subsequently patients will start maintenance treatment during 24 months. Therefore, the total duration of the treatment will be approximately 36 months.

DETAILED DESCRIPTION:
This clinical trial is a multicenter Phase II study designed to evaluate the efficacy and toxicity of an intensive therapeutic approach in 90 patients with asymptomatic high risk multiple myeloma (SMM).

1. - Patients will receive an induction treatment consisting of 6 cycles of carfilzomib, lenalidomide and low-dose dexamethasone (KRd): patients will receive carfilzomib 20-36 mg/m2 IV on days 1, 2, 8, 9, 15 and 16; with oral lenalidomide 25 mg daily on days 1-21, subsequently there will be a rest period of a week (from day 22 to day 27). Moreover, oral dexamethasone 40mg daily will be administered weekly (days 1, 8, 15 and 22).
2. - Following the induction treatment, patients will receive high-dose (200 mg/m2) melphalan-based treatment administered via the intravenous route followed by peripheral blood stem cell transplantation (HDT-ASCT).
3. - The consolidation treatment will consist of 2 cycles of KRd, with the same doses and scheduled of the induction treatment.
4. - Maintenance treatment: all patients, without progression to symptomatic multiple myeloma or toxicity requiring discontinuation of the trial, will receive maintenance treatment during 24 cycles.

This maintenance treatment comprises the administration of lenalidomide 10mg on days 1-21, followed by a rest period of 1 week, with the weekly administration of dexamethasone 20mg.

Treatment will be administrated until the end of the maintenance, although patients will continue in the trial.

If biological progression is observed following the discontinuation of the treatment, lenalidomide and dexamethasone will be reinstituted in order to control the disease again. Lenalidomide 10 mg will be administrated on days 1-21 combined with dexamethasone 20mg on days 1, 8, 15 and 22. All patients will be monitored for asymptomatic disease progression and to collect data regarding on overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* In the investigator's opinion, the patient must be able to fulfill all the clinical trial requirements.
* The patient must voluntarily sign the informed consent before any study procedure that is not part of the standard of care for these patients is performed, with the patient's knowledge that he/she may withdraw from the study at any time, without prejudice to his/her future care.
* The patient must be aged between 18 and 70 years, and eligible to receive high-dose therapy and autologous peripheral blood stem cell transplant.
* The patient must be diagnosed with smoldering multiple myeloma at high risk of progressing to symptomatic multiple myeloma, or at ultra high risk of progression to symptomatic disease, defined by:
* smoldering multiple myeloma at high risk of progression to symptomatic disease:

Bone marrow infiltration with plasma cells (PCs) greater than or equal 10% and presence of a monoclonal component, immunoglobulin G (IgG) greater than3 g/dL or IgA greater than 2 g/dL or Bence Jones proteinuria greater than 1 g/24h and absence of lytic lesions, hypercalcemia, renal failure (creatinine less than 2 mg/dL) and anemia (hemoglobin greater than 10 gr/dL or not 2 gr/dL below the lower limit of normal).

Bone marrow infiltration with PCs greater than or equal 10% OR IgG greater than 3 g/dL or immunoglobulin A (IgA) greater than 2 g/dL or Bence Jones proteinuria greater than 1g/24h (but not both together) and always in the absence of lytic lesions, hypercalcemia, renal failure and anemia. These patients may be included in the study if they meet the following additional criteria: A percentage of phenotypically aberrant plasma cells (PCs) within the bone marrow (BM) PC compartment (aPC/ BM PC) greater than or equal 95% and immunoapheresis, defined as a reduction in the levels of 1 or 2 immunoglobulin (Igs) of more than 25% compared with the normal values of the corresponding Ig.

- smoldering multiple myeloma at ultra high risk of progression to symptomatic disease:

Presence of more than 1 focal lesion in MRI (ideally whole body MRI).

Infiltration in the BM equal or higher than 60%.

Ratio of involved/uninvolved serum Friend leukemia cell (FLC) higher than 100.

* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status less than 2.
* The patient must be able to attend the scheduled visits.
* Women of childbearing potential must have a negative pregnancy test (serum or urine) within the 14 days before the starting the study drug. In addition, sexually active women must agree to use contraceptive methods (hormone contraceptives [oral, injectable or implanted], tubal ligation, intrauterine device, barrier contraceptives with spermicide or have a vasectomised partner) while receiving the study drug. Women of childbearing potential must agree to undergo pregnancy tests every 4 weeks while receiving the study drug (every 14 days for women with irregular menstrual cycles) and 4 weeks after the last dose of study drug.

Exclusion Criteria:

* Any physical condition or psychiatric disorder that would prevent the patient from signing or understanding the informed consent form.
* Previous treatment for smoldering multiple myeloma.
* Pregnancy or breastfeeding.
* Presence of lytic lesions, anemia, renal failure or hypercalcemia.
* Any of the following laboratory abnormalities:

Absolute neutrophil count (ANC) less than 1,000/mm3

Platelet count less than 75,000/mm3.

Serum GOT or glutamic pyruvic transaminase (GPT) greater than 3 x upper limit of normal

Serum total bilirubin greater than 2 x upper limit of normal

* Prior history of neoplasm other than multiple myeloma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the patient has been disease-free for > 5 years.
* Major surgery within 4 weeks before inclusion in the study.
* Known active infection by human acquired immunodeficiency virus, B or C hepatitis virus.
* Any investigational drug within 30 days before inclusion in the study.
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to enrolment.
* Unstable angina or myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
* Uncontrolled hypertension or uncontrolled diabetes.
* Significant neuropathy (Grades 3?4, or Grade 2 with pain) within 14 days prior to enrollment.
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib).
* Contraindication to any of the required concomitant drugs or supportive treatments, including intolerance to hydration due to pre-existing pulmonary or cardiac impairment.
* Left ventricular ejection fraction (LVEF) less than 40
* Pulmonary hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy- Number of Immunophenotypic complete remission rate (Flow-CR) at day +100 after induction and HDT-ASCT | 4 months
  Number of Immunophenotypic complete remission rate (Flow-CR) at day +100 after induction and HDT-ASCT

SECONDARY OUTCOMES:
Efficacy - Number of Response rates after the different parts of the treatment, induction, HDT-ASCT, consolidation and maintenance | up to 24 weeks
  Number of Response rates after the different parts of the treatment, induction, HDT-ASCT, consolidation and maintenance
Efficacy- Months to progression free survival | 60 months
  Months to progression free survival
Efficacy -Months to overall survival | 60 months
  Months to overall survival
Relapse or progression patterns in the group of patients requiring a rescue therapy after june 2020. | Up to 84 months (from june 2020)
  Relapse or progression patterns after first line treatment with KRd->PBPCT->KRd->Rd, in the group of patients requiring a rescue therapy after june 2020.
Response rate of rescue therapy in the group of patients requiring a rescue therapy after june 2020. | Up to 84 months (from june 2020)
  Response rate achieved with daratumumab, pomalidomide and dexamethasone (DPd) as rescue therapy, by evaluating all response categories, including immunophenotypic response, sCR, CR, VGPR, PR and SD.
Progression Free Survival (PFS) and Overall Survival (OS) from the date of relapse / progression of disease | Up to 84 months (from june 2020)
  PFS and OS from the date of relapse / progression of disease, in the group of patients requiring a rescue therapy.
Biological studies in the group of patients requiring a rescue therapy. | Up to 84 months (from june 2020)
  Phenotypic and molecular assessment of the tumor clone that appears in the moment of relapse or disease progression (DP), and comparison against the tumor clone characterized at the moment of inclusion in the first part of the trial.
Study of patient immune profile in the group of patients requiring a rescue therapy. | Up to 84 months (from june 2020)
  Assessment of patient immune profile at the moment of inclusion in this modification, and assessment of evolution under DPd treatment.
Study of patient immune profile depending on type of relapse, in the group of patients requiring a rescue therapy. | Up to 84 months (from june 2020)
  Assessment of immune profile at the moment of inclusion in patients in biochemical relapse vs. those in symptomatic relapse.

CONTACTS AND LOCATIONS:
Locations (16):
- Spain (16):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Clínica Universidad de Navarra, Pamplona
  - Hospital de Son Llàtzer, Plama de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Reina Sofía, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Mateos MV, Martinez-Lopez J, Rodriguez Otero P, Gonzalez-Calle V, Gonzalez MS, Oriol A, Gutierrez NC, Rios-Tamayo R, Rosinol L, Alvarez Rivas MA, Bargay J, Gonzalez-Rodriguez AP, Alegre A, Escalante F, Inigo Rodriguez MB, De La Rubia J, Teruel AI, de Arriba F, Palomera L, Hernandez MT, Lopez Jimenez J, Reinoso-Segura M, Garcia Mateo A, Ocio EM, Paiva B, Puig N, Cedena MT, Blade J, Lahuerta JJ, San-Miguel JF; Spanish Myeloma Group (GEM-Pethema). Curative Strategy for High-Risk Smoldering Myeloma: Carfilzomib, Lenalidomide, and Dexamethasone (KRd) Followed by Transplant, KRd Consolidation, and Rd Maintenance. J Clin Oncol. 2024 Sep 20;42(27):3247-3256. doi: 10.1200/JCO.23.02771. Epub 2024 Jul 22. PMID 39038268